CLINICAL TRIAL: NCT05287490
Title: Clinical Evaluation of Combined Treatment With Bi-Polar Radio-Frequency and Electrical Muscle Stimulation for Symptoms of Mixed Urinary Incontinence (MUI)
Brief Title: Bi-Polar Radio-Frequency and Electrical Muscle Stimulation for Symptoms of Mixed Urinary Incontinence (MUI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO609893A
Record Dates: First submitted 2022-02-15; First posted 2022-03-18 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-02

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- treatment (Experimental)
  Interventions: Device: FormaV and VTone

INTERVENTIONS:
Device: FormaV and VTone — Eligible subjects will receive 3 treatments(every 2 weeks) with the FormaV and VTone Applicators according to the study protocol.

SUMMARY:
The objective of this trial is to evaluate the safety and efficacy of the combined FormaV and VTone Applicators for Symptoms of Mixed Urinary Incontinence.

Eligible subjects will receive 3 treatments(every 2 weeks) with the FormaV and VTone Applicators according to the study protocol.

The subject will return for 3 follow-up visits: 4 weeks (1M FU), 3 months follow up (3M FU), 6 months follow up (6M FU) after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.
* Female subjects, 20 to 75 years of age at the time of enrolment with moderate to severe symptoms of MUI, who had scored a relative even proportion of urge and stress subscale scores on the Medical, Epidemiologic, and Social Aspects of Aging Urinary Incontinence (MESA) Questionnaire completed at the screening assessment
* General good health confirmed by medical history and examination of the treated area.
* The patients should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other aesthetic treatment methods for the last 6 months and during the entire study period.

Exclusion Criteria:

7.5 Exclusion criteria

* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
* Patients who have vaginal metal piercing, or intrauterine contraceptive device (IUCD or ICD or coil or any other device made of metal).
* Permanent implant in the treated area such as metal plates and screws, silicone implants or an injected chemical substance, unless deep enough in the periostal plane.
* Current or history of cancer, or premalignant condition in the treatment area.
* Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy and nursing.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* History of bleeding coagulopathies or use of anticoagulants in the last 10 days.
* Any surgery in treated area within 3 months prior to treatment.
* Simultaneous participation in another investigator drug or device study or completion of the follow-up phase for the primary endpoint of any previous study less than 30 days prior to the first evaluation in this study.
* Six months delay is required if other recent treatments like light, CO2 laser or RF were performed on the same area.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* Simultaneously participating in another investigator drug or device study or has completed the follow-up phase for the primary endpoint of any previous study less than 30 days prior to the first evaluation in this study.
* As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the patient

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Cough stress test | Baseline through month 6
  Change as measured by standardized cough stress test performed in standing position before treatment and 6 months after the treatment
Quality of Life (IQOL) Questionnaire | baseline through month 6
  The effect of the treatment on urinary symptoms and quality of life by means of the Incontinence Quality of Life (IQOL) Questionnaire.
Female Sexual Function Index questionnaire | baseline through month 6
  The effect of the treatment on female sexual function by means of Female Sexual Function Index
Urogenital Distress Inventory 6 Questionnaire | baseline through month 6
  The effect of the treatment on urinary symptoms by means of Urogenital Distress Inventory 6 Questionnaire
Medical, Epidemiologic, and Social Aspects of Aging Urinary Incontinence (MESA) Questionnaire | baseline through month 6
  The effect of the treatment on urinary symptoms by means of Medical, Epidemiologic, and Social Aspects of Aging Urinary Incontinence (MESA) Questionnaire (
Patient Global Impression of Improvement (PGI), using a 5-point Likert scale | month 6
  The rate of satisfaction of patients with treatment assessed by the Patient Global Impression of Improvement (PGI), using a 5-point Likert scale

SECONDARY OUTCOMES:
Discomfort scale | post treatment
  A 10cm visual analog scale from 0 (no discomfort) to 10 (worst possible discomfort) to measure discomfort associated with probe insertion, and RF/EMS energy application at the treatment visit
Adverse events | throughout the study
  Number, severity and type of any adverse event recorded throughout the course of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Advanced Women's Care of the Lowcountry, PC, Bluffton, South Carolina
  - Lisa M Jukes MD, West Lake Hills, Texas

IPD SHARING:
Plan to Share IPD: Undecided